CLINICAL TRIAL: NCT03132103
Title: The Effect of Vitamin D Supplementation on Vitamin D Status, Immunity and Physical Performance
Brief Title: Vitamin D Supplementation and Immunity/Physical Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangor University (Other)
Collaborators: University of East Anglia (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 692/Gen/10
Record Dates: First submitted 2017-03-30; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Vitamin D Status
Keywords: Vitamin D deficiency; Simulated sunlight radiation; Oral vitamin D3
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solar simulated radiation (SSR) (Experimental): Solar simulated radiation (SSR)
  Interventions: Radiation: Solar simulated radiation (SSR)
- Placebo SSR (Placebo Comparator): Placebo SSR
  Interventions: Radiation: Placebo SSR
- Oral Vitamin D3 (Experimental): Oral Vitamin D3
  Interventions: Dietary Supplement: Oral Vitamin D3
- Placebo Oral Vitamin D3 (Placebo Comparator): Placebo Oral Vitamin D3
  Interventions: Dietary Supplement: Placebo Oral Vitamin D3

INTERVENTIONS:
Dietary Supplement: Oral Vitamin D3
  Arms: Oral Vitamin D3
Dietary Supplement: Placebo Oral Vitamin D3
  Arms: Placebo Oral Vitamin D3
Radiation: Solar simulated radiation (SSR)
  Arms: Solar simulated radiation (SSR)
Radiation: Placebo SSR
  Arms: Placebo SSR

SUMMARY:
The purpose of this study is to examine the effect of vitamin D supplementation on vitamin D status, immunity and physical performance.

DETAILED DESCRIPTION:
Vitamin D plays a key role in bone mineralisation and has been linked to immune defence maintenance and muscle function. Vitamin D is primarily obtained from endogenous synthesis in response to skin sunlight exposure and follows a seasonal pattern; whereby, vitamin D levels peak at the end of the summer and fall to a trough during winter. If winter vitamin D levels can be increased to match those found in summer using supplementation, it is proposed sufficient vitamin D levels will improve physical performance and reduce susceptibility to illness in military recruits.

ELIGIBILITY:
Inclusion Criteria:

* Passed medical assessment by medical doctor

Exclusion Criteria:

* Medically deferred by medical doctor
* Regular sun bed use
* Holiday in a hot sunny climate in <3 months
* Regular vitamin D supplementation

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-04-28 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status | Up to 20 months
  Circulating 25-hydroxy-vitamin D, 1,25-d OH(OH)D

SECONDARY OUTCOMES:
Physical performance 1 | Up to 20 months
  Vertical Jump height (cm) and peak power output (watts)
Physical performance 2 | Up to 20 months
  Maximal dynamic lift strength (kg)
Physical performance 3 | Up to 20 months
  Multi-stage fitness test predicted VO2max (mL/kg/min)
Hepatitis B antibody | Up to 20 months
  Antibody produced in response to the presence of Hepatitis B antigen (e.g. Hepatitis B vaccine)
Mucosal immunity | Up to 20 months
  Secretory Immunoglobulin A levels

CONTACTS AND LOCATIONS:
Locations (1):
- Infantry Training Centre, Catterick, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kashi DS, Oliver SJ, Wentz LM, Roberts R, Carswell AT, Tang JCY, Jackson S, Izard RM, Allan D, Rhodes LE, Fraser WD, Greeves JP, Walsh NP. Vitamin D and the hepatitis B vaccine response: a prospective cohort study and a randomized, placebo-controlled oral vitamin D3 and simulated sunlight supplementation trial in healthy adults. Eur J Nutr. 2021 Feb;60(1):475-491. doi: 10.1007/s00394-020-02261-w. Epub 2020 May 10. PMID 32390123